CLINICAL TRIAL: NCT00528970
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study of Intravenous Methylnaltrexone (MOA-728) for the Treatment of Post Operative Ileus After Ventral Hernia Repair
Brief Title: A Study Evaluating Intravenous (IV) MOA-728 for the Treatment of Postoperative Ileus (POI) in Participants After Ventral Hernia Repair
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch Health Americas, Inc. (Industry)
Collaborators: Progenics Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3200L2-301
Record Dates: First submitted 2007-09-11; First posted 2007-09-14 (Estimated); Results first posted 2019-09-04 (Actual); Last update posted 2019-09-04 (Actual); Status verified 2019-08

CONDITIONS: Ileus
Keywords: POI; Hernia; Ventral Wall Hernia Repair; Post Operative Ileus
MeSH Terms: conditions — Ileus; Hernia | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (3):
- MOA-728 12 mg (Experimental): Participants will receive methylnaltrexone (MOA-728) 12 mg as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug will be administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple is placed in the participant). Dose administration will be continued for a maximum of 10 days.
  Interventions: Drug: MOA-728
- MOA-728 24 mg (Experimental): Participants will receive MOA-728 24 mg as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug will be administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple is placed in the participant). Dose administration will be continued for a maximum of 10 days.
  Interventions: Drug: MOA-728
- Placebo (Placebo Comparator): Participants will receive placebo matching to MOA-728 as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug will be administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple is placed in the participant). Dose administration will be continued for a maximum of 10 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MOA-728 — MOA-728 will be administered per the dose and schedule specified in the arm.
  Other Names: Methylnaltrexone
  Arms: MOA-728 12 mg; MOA-728 24 mg
Drug: Placebo — Placebo matching to MOA-728 will be administered per the schedule specified in the arm.
  Arms: Placebo

SUMMARY:
This study will evaluate the safety and efficacy of two different dose regimens (12 milligrams [mg] and 24 mg) of IV MOA-728 versus placebo in shortening the time to return of bowel function in participants receiving opioid analgesia administered via patient-controlled anesthesia (PCA), and who had undergone repair of large (greater than or equal to [≥]10 centimeters) ventral hernias with or without a mesh prosthesis via laparotomy or laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Males and females, ages 18 and older.
* Scheduled for ventral wall hernia repair with general anesthesia.
* Meets the American Society of Anesthesiologists physical status I, II, or III.

Exclusion Criteria:

* Received investigational drug or procedure within 30 days of randomization.
* Women who are pregnant or lactating.
* Calculated creatinine clearance (Cockcroft-Gault glomerular filtration rate [GFR] formula) less than or equal to (</=) 50 milliliters/minute (mL/min).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Actual)
Dates: Start 2007-10-17 (Actual); Primary Completion 2008-02-05 (Actual); Study Completion 2008-02-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lindsey Mathew, Study Director — Bausch Health Americas, Inc.
Locations (95):
- United States (65):
  - Benton, Arkansas
  - Colton, California
  - Laguna Hills, California
  - Loma Linda, California
  - Long Beach, California
  - Los Angeles, California
  - Orange, California
  - San Jose, California
  - Santa Barbara, California
  - Denver, Colorado
  - Inverness, Florida
  - Jacksonville, Florida
  - Melbourne, Florida
  - Miami, Florida
  - Naples, Florida
  - Orlando, Florida
  - Pensacola, Florida
  - Tampa, Florida
  - Peoria, Illinois
  - Des Moines, Iowa
  - Kansas City, Kansas
  - Lexington, Kentucky
  - Baltimore, Maryland
  - Boston, Massachusetts
  - Springfield, Massachusetts
  - Ann Arbor, Michigan
  - Detroit, Michigan
  - Flint, Michigan
  - Jackson, Mississippi
  - Columbia, Missouri
  - Omaha, Nebraska
  - New Brunswick, New Jersey
  - Albuquerque, New Mexico
  - Albany, New York
  - New York, New York
  - Stony Brook, New York
  - Syracuse, New York
  - The Bronx, New York
  - Chapel Hill, North Carolina
  - Durham, North Carolina
  - Winston-Salem, North Carolina
  - Cincinnati, Ohio
  - Cleveland, Ohio
  - Columbus, Ohio
  - Oklahoma City, Oklahoma
  - Bend, Oregon
  - Portland, Oregon
  - Hershey, Pennsylvania
  - Philadelphia, Pennsylvania
  - Pittsburgh, Pennsylvania
  - Sellersville, Pennsylvania
  - Providence, Rhode Island
  - Sioux Falls, South Dakota
  - Knoxville, Tennessee
  - Memphis, Tennessee
  - Nashville, Tennessee
  - Fort Worth, Texas
  - San Antonio, Texas
  - Temple, Texas
  - Norfolk, Virginia
  - Winchester, Virginia
  - Bellevue, Washington
  - Tacoma, Washington
  - Morgantown, West Virginia
  - Milwaukee, Wisconsin
- Australia (2):
  - Adelaide SA
  - Elizabeth Vale SA
- Belgium (2):
  - Wilrijkstraat 10, Edegem
  - De Pintelaan 185, Gent Belgium
- Canada (3):
  - Edmonton, Alberta
  - Vancouver, British Columbia
  - Montreal, Quebec
- Germany (3):
  - Nussbaumstrasse 20, Muenchen
  - Augustenburger Platz 1, State of Berlin
  - Heidelberg
- Hungary (4):
  - Nyíregyháza
  - Pécs
  - Székesfehérvár
  - Veszprém
- Italy (4):
  - Corso Giovecca 203, Ferrara
  - Gemelli, Rome
  - Padua, Via Giustiniani 2
  - Bergamo
- Netherlands (2):
  - Jan Toorpstraat 164, Amsterdam
  - Roosendaal
- Poland (3):
  - Powstancow Wielkopolskich 72, Szczecin
  - Bydgoszcz
  - Polnocna 42, Łódź Voivodeship
- South Africa (6):
  - Durban Kwa-Zulu, KwaZulu-Natal
  - Somerset West, Western Cape
  - Worcester, Western Cape
  - Moreletapark Pretoria
  - Pretoria
  - Pretoria Gauteng
- Kangnam-Gu, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Postoperative participants (who had undergone repair of large [at least 10 centimeters] ventral hernias, with or without mesh prosthesis via laparotomy or laparoscopy) were randomized in 1:1:1 ratio to either MOA-728 24 mg, MOA-728 12 mg, or placebo treatment groups.
Pre-assignment Details: Participants were prospectively stratified by type of surgery (laparotomy or laparoscopy) and geographic region.
Groups:
- MOA-728 12 mg: Participants received methylnaltrexone (MOA-728) 12 milligrams (mg) as an intravenous (IV) infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug was administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple was placed in the participant). Dose administration was continued for a maximum of 10 days.
- MOA-728 24 mg: Participants received MOA-728 24 mg as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug was administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple was placed in the participant). Dose administration was continued for a maximum of 10 days.
- Placebo: Participants received placebo matched to MOA-728 as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug was administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple was placed in the participant). Dose administration was continued for a maximum of 10 days.
Period: Overall Study
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Started | 124 | 125 | 125
Received at Least 1 Dose of Study Drug (Modified intent-to-treat (mITT)/Safety population) | 124 | 125 | 124
Completed | 110 | 110 | 105
Not Completed | 14 | 15 | 20
Not completed — Adverse Event | 6 | 8 | 5
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Other than specified | 2 | 3 | 3
Not completed — Protocol Violation | 2 | 1 | 4
Not completed — Lack of Efficacy | 0 | 0 | 1
Not completed — Withdrawal by Subject | 4 | 3 | 5
Not completed — Randomized but not treated | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all randomized participants who received at least 1 dose of study drug.
Groups:
- MOA-728 12 mg: Participants received MOA-728 12 mg as an IV infusion over approximately 20 minutes for approximately every 6 hours for a total of 4 doses in 24-hour period. The first dose of study drug was administered within approximately 90 minutes after completion of the surgical procedure (defined as the time when the last skin suture or staple was placed in the participant). Dose administration was continued for a maximum of 10 days.
- Total: Total of all reporting groups
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo | Total
Number analyzed (Participants) | 124 | 125 | 124 | 373
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.11 (13.25) | 55.21 (13.05) | 55.82 (13.52) | 56.05 (13.26)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 63 | 66 | 68 | 197
  Male | 61 | 59 | 56 | 176

OUTCOME MEASURES:

1. Primary Outcome: Time to First Bowel Movement
Description: Time to first bowel movement was measured from the end of surgery (defined as the time when the last skin suture or staple was placed in the participant). Time of the first bowel movement was recorded on the electronic case report form (eCRF). The first bowel movement was defined as a normal stool for a postoperative participant based on the clinical judgment of the investigator or designee. Analysis was performed by Kaplan-Meier estimate. Participants who had a bowel movement but were readmitted to the hospital within 1 week after discharge with a diagnosis of postoperative ileus (POI) were considered censored at the time of the first bowel movement as if the bowel movement had not occurred.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: hours
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Number analyzed (Participants) | 124 | 125 | 124
hours | 93.3 (3.2) | 100.4 (4.2) | 91.3 (3.9)
Statistical Analysis 1: Comparison: MOA-728 12 mg vs Placebo; Analysis was performed using log-rank test stratified by surgery type and region for comparisons of survival distributions for active MOA versus Placebo group; Test type: Other; p = 0.944, Log Rank — Threshold for significance at 0.05 level; Mean Difference (Final Values) = 2.0
Statistical Analysis 2: Comparison: MOA-728 24 mg vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other; p = 0.208, Log Rank — Threshold for significance at 0.05 level; Mean Difference (Final Values) = 9.1

2. Secondary Outcome: Time to Discharge Eligibility
Description: Time to discharge eligibility was measured from the end of surgery (defined as the time when the last skin suture or staple was placed in the participant). Discharge eligibility was defined as tolerance of oral intake of liquids greater than (>) 500 milliliters (mL) per 8 hours without nausea or retching/vomiting. Analysis was performed by Kaplan-Meier estimate.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: hours
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Number analyzed (Participants) | 124 | 125 | 124
hours | 44.9 (2.9) | 51.4 (5.1) | 41.4 (3.4)

3. Secondary Outcome: Time to Discharge Order Written From the End of Surgery
Description: The investigator or designee recorded the time of the order. Participants re-admitted to the hospital with a diagnosis of POI within 7 days after discharge was considered treatment failures. Analysis was performed by Kaplan-Meier estimate.
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 10
Population: mITT population included all randomized participants who received at least 1 dose of study drug.
Measure: Mean (Standard Error); unit: hours
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Number analyzed (Participants) | 124 | 125 | 124
hours | 130.6 (15.52) | 123.8 (6.8) | 132.9 (14.1)

4. Secondary Outcome: Number of Participants With Clinically Meaningful Events (CMEs) for Nausea or Retching/Vomiting at Day 2 (24 Hours) as Evaluated by the Opioid-Related Symptom Distress Scale (SDS)
Description: CMEs were defined using opioid-related SDS (assessed participant-reported levels of severity concerning 10 symptoms associated with opioid medication usage: fatigue, drowsiness, inability to concentrate, nausea, dizziness, constipation, itching, difficulty with urination, confusion and retching/vomiting). CME = any symptom rated as severe (3) or very severe (4), with the exception of confusion. A total CME score was calculated by summing the number of CMEs across symptoms and ranged from 0 to 9. CME was counted for either nausea or vomiting/retching, or both and reported in this outcome measure.
Time Frame: Day 2
Population: mITT population included all randomized participants who received at least 1 dose of study drug. Here, 'Overall number of participants analyzed' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Number analyzed (Participants) | 115 | 113 | 113
Participants | 10 | 19 | 7

ADVERSE EVENTS:
Time Frame: Day 1 (From the time of end of surgery [that is; from the first dose of study drug administration]) up to Day 15
Description: Safety population included all randomized participants who received at least 1 dose of study drug.
Arm/Group | MOA-728 12 mg | MOA-728 24 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 20/124 | 17/125 | 28/124
Other Adverse Events (participants affected / at risk) | 68/124 | 71/125 | 73/124
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MOA-728 12 mg (N=124) | MOA-728 24 mg (N=125) | Placebo (N=124)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 2
Coagulopathy (Blood and lymphatic system disorders) | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1 | 1
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Abdominal wall haematoma (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Enterocutaneous fistula (Gastrointestinal disorders) | 0 | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 0 | 1
Intestinal fistula (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0
Localised intraabdominal fluid collection (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 0 | 1
Hernia (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 0 | 0
Wound necrosis (General disorders) | 0 | 1 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 0 | 1
Bacteraemia (Infections and infestations) | 0 | 1 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 1 | 0 | 0
Incision site infection (Infections and infestations) | 1 | 0 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0
Post procedural infection (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Wound infection (Infections and infestations) | 5 | 0 | 2
Wound infection staphylococcal (Infections and infestations) | 1 | 2 | 0
Incisional hernia, obstructive (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 3 | 1 | 2
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 0 | 1 | 2
Wound dehiscence (Injury, poisoning and procedural complications) | 0 | 0 | 3
Wound secretion (Injury, poisoning and procedural complications) | 1 | 0 | 1
Liver function test abnormal (Investigations) | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin necrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MOA-728 12 mg (N=124) | MOA-728 24 mg (N=125) | Placebo (N=124)
Tachycardia (Cardiac disorders) | 4 | 2 | 8
Constipation (Gastrointestinal disorders) | 10 | 13 | 11
Nausea (Gastrointestinal disorders) | 39 | 33 | 38
Vomiting (Gastrointestinal disorders) | 16 | 20 | 21
Fatigue (General disorders) | 7 | 1 | 3
Pyrexia (General disorders) | 17 | 15 | 18
Hypokalaemia (Metabolism and nutrition disorders) | 4 | 10 | 4
Dizziness (Nervous system disorders) | 7 | 4 | 5
Headache (Nervous system disorders) | 8 | 9 | 13
Somnolence (Nervous system disorders) | 7 | 1 | 6
Urinary retention (Renal and urinary disorders) | 12 | 10 | 11
Pruritus (Skin and subcutaneous tissue disorders) | 17 | 11 | 17
Hypertension (Vascular disorders) | 4 | 8 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Please contact Sponsor directly for additional information.